CLINICAL TRIAL: NCT04199416
Title: Effectiveness of an Interactive, Multi-functional Mobile App-based Technology in Endogenous Healthcare for Individuals With or at Risk of Knee Osteoarthritis: A 12-month Randomized Controlled Trial
Brief Title: Effectiveness of a Mobile App for Individuals With or at Risk of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Calvin Or, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HMRF 17181291
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Knee Pain/Osteoarthritis; Digital Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mRehab app (Experimental): Participants randomized to the intervention group will be given the mRehab app free of charge to perform self-management of their knees in their homes.
  Interventions: Device: mRehab app
- Sham app (Sham Comparator): Participants randomized to the control group will receive a sham app free of charge to perform self-management of their knees in their homes.
  Interventions: Device: Sham app

INTERVENTIONS:
Device: mRehab app — The mRehab app will be an interactive system with a user-friendly graphical user interface to provide multiple motivational functions that engage individuals in their prescribed home exercises. The app will contain video-based lower limb strengthening and aerobic exercise materials, health information, and motivational functions to increase their access to rehabilitation and care resources to augment their self-management ability.
  Arms: mRehab app
Device: Sham app — The sham app will only contain educational components and text-based exercise recommendations.
  Arms: Sham app

SUMMARY:
To develop and examine an interactive, multi-functional mobile app-based technology designed to encourage endogenous health care using a 12-month randomized controlled trial to demonstrate whether knee osteoarthritis (KOA)-at-risk individuals and KOA-diagnosed patients can improve their knee pain, physical function, and other relevant outcomes by using the technology to support knee/KOA self-management.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA), the most common degenerative condition affecting the peripheral weight-bearing joints, leads to pain, restricted mobility, and financial and moral burden. These effects will increase with rising numbers of incidents, exacerbated by population aging and obesity. Zhang et al. found KOA in 43% and 22% (15% and 6% in symptomatic individuals) of Chinese women and men, respectively, 60 years or older. In the United States, KOA affects 12% of the elderly population, and it is projected that the need for total knee replacement (TKR) to treat end-stage KOA will grow by 673% to 3.48 million procedures a year from 2005 to 2030, with the demand for TKR revision doubling from 2005 to 2015. Hong Kong's public hospitals performed 6658 TKRs from 2011 to 2014, with 10,000 cases wait-listed for 2016. These figures suggest that KOA will impose significant and increasing pressure on Hong Kong's healthcare system.

As quadriceps muscle weakness increases the risk of KOA, its symptoms should be alleviated by leg muscle strengthening. Land-based exercise has been effective under close monitoring and supervision. A recent Cochrane Review involving 54 studies concluded that there is moderate to high-quality evidence that land-based exercises significantly improve muscle strength, physical function, and quality of life and reduce pain in KOA patients. The effect of such exercises is comparable to that of nonsteroidal anti-inflammatory drugs with no significant adverse effects. However, therapist-delivered exercise is costly and often impractical, especially in a public-health context, and Internet-delivered exercise regimes represent an alternative approach. In today's information technology (IT)-enabled environment, mobile apps are readily accessible to users of untethered devices (e.g., smartphones). The "any-where, any-time" mobile IT could be exploited to more effectively manage KOA by encouraging self-motivation to substitute for direct monitoring. This study will present "IT-centered endogenous healthcare" as a public policy to boost self-help in primary care and test its practicability and efficacy in KOA management in Hong Kong. The word "endogenous" suggests that self-motivation is a form of self-insurance in primary care. It is further suggested that demand-side incentives will be needed to induce individuals to incrementally allocate more resources (particularly time and effort) to incrementally self-insure health at the primary level.

On the supply side, IT-based healthcare products have been mainly designed for commercial considerations such as marketing and are insufficiently focused on function for purposes of public health and policy. We follow Liao-Cheung's approach to reify demand-side incentives in the form of a publicly funded (and hence free) mobile app, the adoption of which could encourage self-insurance among individuals with knee problems or KOA. The users' time and effort will initially be rewarded by the app's user-friendliness and lack of a fee. The study's technology intervention, "mobile rehabilitation (mRehab) app", will link smartphones to videos of evidence-based, physiotherapist-prescribed exercises to alleviate knee/KOA symptoms, together with educational (e.g., diet and behavioral modifications) and motivational components. This mobile IT platform will have easier and wider accessibility than exercises delivered via tethered devices (e.g., desktop computers), and it can engage the users' interest whenever and wherever KOA effects are felt. Over time, self-motivation is also enhanced by high-frequency prompts, periodic upgrades with feedback, support from Internet KOA-awareness groups, the possibility of accumulating one's own health-data to facilitate queries and dialogue, and (most importantly) monitoring the health progression predicted by the exercise regimen.

A natural research sample follows in the form of IT-enabled individuals with knee/KOA problems. The proposed hypothesis is then offered that sustained use of the mRehab app will significantly reduce the symptoms and improve functions of individuals with quadriceps weakness and knee pain or KOA over time and compared to a sham app (the analytical control). The effectiveness of the mRehab app regarding this hypothesis will be tested in two samples: (1) KOA-at-risk individuals and (2) KOA-diagnosed patients, in a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion criteria for all participants:

* at least 50 years of age,
* a regular smartphone user,
* able to speak Cantonese and read Chinese,
* able to perform the exercises required in the physical assessments,
* able to provide written informed consent.

Inclusion criteria for KOA-at-risk participants:

* with subnormal quadriceps strength (as defined by the inability to complete five repetitions of a sit-to-stand test in less than 8 seconds [50 to 70 years of age], 10 seconds [70 to 79 years of age], or 12 seconds [80 years or older])
* with significant chronic knee pain (i.e., ≥2/10 on the 11-point Numerical Pain Rating Scale for more than 3 months on most days of the previous month, aggravated by weight-bearing or movement)
* without regular medical follow-up for knee problems

Inclusion criteria for KOA-diagnosed participants:

* with symptomatic radiographic KOA and being followed-up in hospitals
* have radiographic evidence of grade 2 to 3 KOA on the Kellgren-Lawrence scale in the posteroanterior and/or skyline view or the presence of lateral/posterior osteophytes.

Exclusion criteria:

* have a cognitive impairment,
* have nonambulatory status,
* have systemic inflammatory arthritis (e.g., gout),
* have a history of knee or hip replacement surgery,
* have a history of trauma or surgical arthroscopy of either knee within the past 6 months,
* involve in a similar study,
* participate in a knee exercise program within the past 6 months,
* have an intra-articular injection to the knee within the past 3 months,
* have recent or imminent surgery (within 3 months),
* have medical co-morbidities that preclude participation in exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in knee pain | from baseline to 3, 6, 9, and 12 months
  Knee pain will be assessed on a 11-point Numerical Pain Rating Scale, with 0 representing no pain and 10 representing the worst possible pain.
Changes in physical function of the knee | from baseline to 3, 6, 9, and 12 months
  Physical function will be measured with the 17-item physical function for daily living subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS). A 5-point Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems).

SECONDARY OUTCOMES:
Changes in lower limb function | from baseline to 3, 6, 9, and 12 months
  Lower limb function will be assessed by a 40-m fast-paced walking test, a 9-step stair-climb test, a five-repetition sit-to-stand test, active and passive ranges of motion of the hip and knee joints, and the mini-balance evaluation system test (mini-BESTest).
Changes in lower limb muscle strength | from baseline to 3, 6, 9, and 12 months
  Maximal isometric strength of the quadriceps and hamstrings will be assessed by a handheld dynamometer.
Changes in health-related physical activity | from baseline to 3, 6, 9, and 12 months
  Health-related physical activity will be assessed using the Chinese version of international physical activity questionnaire. This questionnaire asks participants to report the frequency and duration of walking, all vigorous and moderate activities lasting at least 10 min, plus time spent in sedentary activity (sitting and lying awake) during the past 7 days. The data were converted to metabolic equivalent scores for each type of activity, with higher score indicating more physical activity.
Changes in self-efficacy for coping with knee problems | from baseline to 3, 6, 9, and 12 months
  Self-efficacy will be assessed using a 5-item self-efficacy scale modified from an existing validated scale, with scores ranging from 1 (not at all confident) to 10 (totally confident).
Changes in health-related quality of life | from baseline to 3, 6, 9, and 12 months
  Health-related quality of life will be measured using the Chinese version of the EuroQoL 5-dimension 5-level (EQ-5D-5L) questionnaire, which consists of the EuroQoL 5-dimension (EQ-5D) descriptive system and the EQ visual analogue scale (VAS). The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension is rated on a 3-point scale (i.e., no problems, some problems, and extreme problems). The EQ VAS asks the subject to indicate his or her health state on a vertical, visual analog scale with end points of 0 (worst imaginable health state) and 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Hong Kong East Cluster, Hospital Authority, Hong Kong
  - Hong Kong West Cluster, Hospital Authority, Hong Kong
  - New Territories East Cluster, Hospital Authority, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Zhang Y, Xu L, Nevitt MC, Aliabadi P, Yu W, Qin M, Lui LY, Felson DT. Comparison of the prevalence of knee osteoarthritis between the elderly Chinese population in Beijing and whites in the United States: The Beijing Osteoarthritis Study. Arthritis Rheum. 2001 Sep;44(9):2065-71. doi: 10.1002/1529-0131(200109)44:93.0.CO;2-Z. PMID 11592368
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Lee QJ, Mak WP, Wong YC. Mortality following primary total knee replacement in public hospitals in Hong Kong. Hong Kong Med J. 2016 Jun;22(3):237-41. doi: 10.12809/hkmj154712. Epub 2016 May 6. PMID 27149975
- [Background] Oiestad BE, Juhl CB, Eitzen I, Thorlund JB. Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Feb;23(2):171-7. doi: 10.1016/j.joca.2014.10.008. Epub 2014 Nov 1. PMID 25450853
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Bennell KL, Nelligan R, Dobson F, Rini C, Keefe F, Kasza J, French S, Bryant C, Dalwood A, Abbott JH, Hinman RS. Effectiveness of an Internet-Delivered Exercise and Pain-Coping Skills Training Intervention for Persons With Chronic Knee Pain: A Randomized Trial. Ann Intern Med. 2017 Apr 4;166(7):453-462. doi: 10.7326/M16-1714. Epub 2017 Feb 21. PMID 28241215
- [Background] Case MA, Burwick HA, Volpp KG, Patel MS. Accuracy of smartphone applications and wearable devices for tracking physical activity data. JAMA. 2015 Feb 10;313(6):625-6. doi: 10.1001/jama.2014.17841. No abstract available. PMID 25668268
- [Background] Yingyongyudha A, Saengsirisuwan V, Panichaporn W, Boonsinsukh R. The Mini-Balance Evaluation Systems Test (Mini-BESTest) Demonstrates Higher Accuracy in Identifying Older Adult Participants With History of Falls Than Do the BESTest, Berg Balance Scale, or Timed Up and Go Test. J Geriatr Phys Ther. 2016 Apr-Jun;39(2):64-70. doi: 10.1519/JPT.0000000000000050. PMID 25794308
- [Background] Bohannon RW, Bubela DJ, Magasi SR, Wang YC, Gershon RC. Sit-to-stand test: Performance and determinants across the age-span. Isokinet Exerc Sci. 2010;18(4):235-240. doi: 10.3233/IES-2010-0389. PMID 25598584
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Or C, Tao D. A 3-Month Randomized Controlled Pilot Trial of a Patient-Centered, Computer-Based Self-Monitoring System for the Care of Type 2 Diabetes Mellitus and Hypertension. J Med Syst. 2016 Apr;40(4):81. doi: 10.1007/s10916-016-0437-1. Epub 2016 Jan 22. PMID 26802011